CLINICAL TRIAL: NCT01074814
Title: A Pilot Study Utilizing Molecular Profiling by IHC, FISH, DNA Microarray, and Reverse Phase Protein Microarray (RPMA) of Patients' Tumors to Find Potential Targets and Select Treatments for Patients With Metastatic Breast Cancer.
Brief Title: Pilot Study Using Molecular Profiling to Find Potential Targets & Select Treatments for Pts With Met br ca
Acronym: Side-Out
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Translational Drug Development (Other)
Collaborators: Side-Out Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SO-BCA-001
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2022-11

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; Molecular profiling
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metastatic Breast Cancer Patients (Other): Blood drawn for molecular profiling
  Interventions: Drug: Approved therapy will be assigned based on molecular profile and RPMA results

INTERVENTIONS:
Drug: Approved therapy will be assigned based on molecular profile and RPMA results — treatment will be assigned based on IHC< FISH, DNA microarray and RPMA results
  Other Names: Approved therapy will be administered based on molecular profile and RPMA results

SUMMARY:
The purpose of this study is to determine the response rate, that is the % of patients with non-progression of their metastatic breast cancer after 4 months on treatment that was selected by molecular testing and proteomics.

DETAILED DESCRIPTION:
To determine the percent of patients with refractory breast cancer where molecular profiling and RPMA-based protein pathway activation analysis of their tumor, can change the clinical course of their disease (i.e. produce a Growth Modulation Index (GMI) ≥1.3). The GMI is calculated as the ratio of Progression-free survival (PFS) under molecular profiling and RPMA analysis selected treatment to the time to progression (TTP) for the most recent regimen the patient has progressed on.

ELIGIBILITY:
Inclusion Criteria:

* Have a life expectancy of greater than 3 months
* metastatic breast cancer, with measurable or evaluable non-measurable disease
* Have progressed on at least 3 prior chemotherapeutic or biological regimens
* Be defined as refractory to the last line of therapy according to the following criteria: Documented disease progression under the last treatment or within two months of the last treatment dosing AND Have received ≥ 30 days of the last treatment AND Have discontinued for progression by RECIST 1.1 criteria
* ≥18 years of age
* ECOG 0-1
* willing to undergo a biopsy or surgical procedure to obtain tissue
* Must have been off their prior regimen for ≥ 3 weeks or 5 x half life of drug
* Have adequate organ and bone marrow function as defined below:
* Female patients of child-bearing potential must have a negative pregnancy test and agree to use at least one form of contraception during the study and for at least one month after treatment discontinuation. For the purposes of this study, child-bearing potential is defined as: all female patients unless they are post-menopausal for at least one year or are surgically sterile
* Male patients must use a form of barrier contraception approved by the Investigator during the study and for at least one month after treatment discontinuation.

Exclusion Criteria:

* Tumor biopsy intended for use in the current study which was performed more than 2 months prior
* Frozen material is not available/obtained
* Metastatic lesion is not accessible to biopsy
* Patients with > 6 months treatment under the last line of therapy
* Patients with symptomatic CNS metastasis. Patients with a history of CNS metastases who have been treated must be stable without symptoms for 4 weeks after completion of treatment, with image documentation required, and must be either off steroids or on a stable dose of steroids for ≥ 2 weeks prior to enrollment
* Any previous history of another malignancy (other than cured basal cell carcinoma of the skin or cured in-situ carcinoma of the cervix) within 5 years of study entry
* Uncontrolled concurrent illness including, but not limited to, ongoing or active serious infection, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmias, psychiatric illness, or situations that would limit compliance with the study requirements or the ability to willingly give written informed consent
* Known HIV, HBV, HCV infection
* Pregnant or breast-feeding patients or any patient with childbearing potential not using adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gayle Jameson, RNMSNACNP-BC, Principal Investigator — Scottsdale Healthcare
Locations (3):
- United States (3):
  - Tgen Clinical Research Services, Scottsdale, Arizona
  - Fairfax North Virginia Hematology Oncology, Fairfax, Virginia
  - Evergreen Hematology and Oncology, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jameson GS, Petricoin EF, Sachdev J, Liotta LA, Loesch DM, Anthony SP, Chadha MK, Wulfkuhle JD, Gallagher RI, Reeder KA, Pierobon M, Fulk MR, Cantafio NA, Dunetz B, Mikrut WD, Von Hoff DD, Robert NJ. A pilot study utilizing multi-omic molecular profiling to find potential targets and select individualized treatments for patients with previously treated metastatic breast cancer. Breast Cancer Res Treat. 2014 Oct;147(3):579-88. doi: 10.1007/s10549-014-3117-1. Epub 2014 Sep 11. PMID 25209003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The open-label multicenter pilot study accrued patients between March 2010 and June 2012. Three Oncology Practices contributed patients to the study.
Groups:
- Metastatic Breast Cancer Patients: Intervention Details:
  Drug: (will be assigned based on molecular profile and RPMA)
  treatment will be assigned based on IHC< FISH, DNA microarray and RPMA results
Period: Overall Study
Arm/Group | Metastatic Breast Cancer Patients
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Intervention Details:
  Drug: (will be assigned based on molecular profile and RPMA)
  treatment will be assigned based on IHC< FISH, DNA microarray and RPMA results
Arm/Group | Intervention
Number analyzed (Participants) | 25
Age, Customized [Median (Full Range); unit: years]
  age | 58 [33 to 77]
Sex/Gender, Customized [Number; unit: participants]
  Female | 25
Race/Ethnicity, Customized [Number; unit: Participants] — Participants
  Participants
    Asian | 1
    White | 23
    Unknown | 1
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Growth Modulation Index (GMI) Greater Than or Equal to 1.3
Description: The primary objective was to determine the % of patients with refractory breast cancer where MMP-informed selection of approved cancer therapies could change the clinical course of their disease to produce a Growth Modulation Index (GMI) greater than 1.3. The GMI was calculated as the PFS with MMP-selected therapy/time to progression (TTP) on last prior therapy. A GMI of 1.3 was selected because 30% or greater improvement in PFS with MMP-selected therapy compared to previous TTP would be considered clinically meaningful.
Time Frame: 6-20 weeks
Population: A total of 28 patients were enrolled and underwent tumor biopsy for the purposes of this study. 25/28 patients were treated on study with the MMP-selected treatment and were evaluable for the primary end point of GMI.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 25
Participants | 25
Statistical Analysis 1: Comparison: Intervention; Test type: Other; Results for the primary objective - evaluation of GMI - were presented with descriptive statistics as the ration of PFS on current therapy over the PFS on latest therapy. The percentage of patients with GMI greater than 1.3 was displayed along with its corresponding 95% exact confidence interval

ADVERSE EVENTS:
Time Frame: adverse events grade 3 and 4 were collected for 2 years.
Description: The study is a molecular profiling study only. No research intervention.
Groups:
- Intervention: Intervention Details:
  Drug: (will be assigned based on molecular profile and RPMA)
  Basis for decision making:
  treatment will be assigned based on IHC< FISH, DNA microarray and RPMA results
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 5/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=25)
hand-foot syndrome (Skin and subcutaneous tissue disorders) | 3 (3)
vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less